CLINICAL TRIAL: NCT05632536
Title: Comparison of Analgesic Efficacy of Sacral erectOR Spinae Plane Block and Caudal Block in Patients Undergoing Hypospadias Surgery
Brief Title: Comparison of Analgesic Efficacy of ESP Block and Caudal Block in Patients Undergoing Hypospadias Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sevgi Kesici, MD, Associate Professor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 240819
Record Dates: First submitted 2022-10-24; First posted 2022-11-30 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Post Operative Pain; Hypospadias
Keywords: sacral erector spinae plane block; caudal block; hypospadias; pediatric surgery
MeSH Terms: conditions — Pain, Postoperative; Hypospadias

STUDY DESIGN:
Intervention Model Description: Our research will be conducted in a single center as a prospective randomized controlled study. It was planned to include 60 patients from the ASA I-II pediatric patient group aged between 6 months and 7 years, who will undergo hypospadias surgery in our hospital between December 2022 and December 2023, and randomization will be done by closed envelope method. Two groups with sacral ESP and caudal block will be formed, each with 30 patients.
Who Masked: Participant, Care Provider
Masking Description: The study was planned to be performed as a double blind. User sacral ESP and caudal block will be administered by an anesthesiologist not responsible for the perioperative and postoperative management of the patients. A second anesthesiologist, who will be in charge of patient monitoring and data recording, will be unaware of the patients' group assignments. Additionally, parents, surgeons, and other personnel involved in the data collection process will be unaware of the group to which the child is assigned. Surgeons will not be present in the operating room while the anesthesiologist administers the block (sacral ESP block or caudal block). All patients will undergo aseptic skin preparation using Betadine. Since bandages will be applied to two points, the actual injection site will not be known.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- GROUP ESP (Active Comparator): Before the operation, under general anesthesia, group ESP (n=30) patients will be blocked with the sacral ESP block method. By giving the lateral decubitus position, the linear ultrasound probe will be placed in the sterilized area longitudinally on the midline of the sacrum. The erector spinae muscle and the sacral medial crest will be visualized. The 22 gauge, 50 mm needle will be advanced in the direction from cranial to caudal to reach the sacral crest. 0.25% bupivacaine from a dose of 1 mL kg-1 will be aspirated and injected every 2 mL under the erector spina muscle at the level of the median sacral crest at the level of the 4th sacral vertebra. (A test dose will be administered with 1 mL of saline.)
  Interventions: Procedure: SACRAL ESP AND CAUDAL BLOCK
- GROUP C (Sham Comparator): Group C (n=30) patients to whom caudal block will be applied will be placed in the lateral decubitus position and the linear ultrasound probe will be placed longitudinally in the sterilized area on the midline of the sacrum. A 2.5 cm 22 gauge needle will be inserted over the back skin of the sacral hiatus (located distal to the sacrum and formed by the two sacral cornua on its lateral edges) at a 90° position. The sacrococcygeal ligament will be crossed, the needle will be oriented approximately 25° and advanced approximately 2 to 3 mm to reach the sacral canal. After entering the sacral hiatus and confirming the location with negative aspiration method, 1 mL kg-1 0.25% bupivacaine will be injected by aspiration every 2 mL (test dose will be administered with 1 mL saline).
  Interventions: Procedure: SACRAL ESP AND CAUDAL BLOCK

INTERVENTIONS:
Procedure: SACRAL ESP AND CAUDAL BLOCK — Application of ultrasound-guided sacral erector spinae plane (ESP) block or ultrasound-guided caudal block with 1mL/kg 0.25% bupivacaine (local anesthetic) to patients

SUMMARY:
The goal of clinical trial is to compare in of analgesic efficacy of sacrale erector spinae plane (ESP) block and caudal block in participants undergoing hypospadias surgery. Investigators will include children between the ages of 6 months and 7 years in the 1st and 2nd categories in the ASA.

In this study, investigators seek answers to the following questions:

Which of the sacral (ESP) block and caudal block applied to participants undergoing hypospadias surgery has higher postoperative analgesic efficiency than the other? Which of the sacral ESP block and caudal block applied to participants undergoing hypospadias surgery is superior in duration of analgesia? After general anesthesia is administered to the participants, one of the 2 blocks will be administered in a randomized manner and the relevant data will be recorded. This research will be conducted in a single center as a prospective randomized controlled study. It was planned to include 60 participnts from the ASA I-II pediatric participants aged between 6 months and 7 years, who will undergo hypospadias surgery between December 2022-December 2023, and randomization will be done by closed envelope method. Two groups with sacral ESP and caudal block will be formed, each with 30 participants.

DETAILED DESCRIPTION:
This study will be conducted as a prospective, randomized controlled trial at a single center between December 2022 and December 2023. Sixty pediatric participants, aged 6 months to 7 years, classified as ASA I-II, who are scheduled for hypospadias surgery, will be included. Participants will be randomized into two groups: ESP block group and caudal block group, with 30 participants in each group. Randomization will be done using a sealed envelope technique based on computer-generated random numbers..

The study was planned to be performed as a double blind. Sacral ESP and caudal block will be administered by an anesthesiologist not responsible for the perioperative and postoperative management of the participants. A second anesthesiologist, who will be in charge of monitoring and data recording, will be unaware of the participants' group assignments. Additionally, parents, surgeons, and other personnel involved in the data collection process will be unaware of the group to which the child is assigned. Surgeons will not be present in the operating room while the anesthesiologist administers the block (sacral ESP block or caudal block). All participants will undergo aseptic skin preparation using Betadine. Since bandages will be applied to two points, the actual injection site will not be known.

The age, height, weight, gender and ASA scores of the participants in both groups will be recorded.

After the participants are taken to the operation table, standard monitoring will be performed. Heart rate (HR), mean arterial pressure (MAP), body temperature, peripheral oxygen saturation (SpO2) will be monitored and all parameters before surgical incision, after surgical incision, before awakening, postoperative 5 and 30 minutes will be recorded.

All participants will be placed in an IV cannula using 8% sevoflurane in 50/50 O2 / air for 2 - 4 minutes with a face mask, followed by induction of inhaled anesthesia. All participants will be placed in I-gel (supraglottic airway vehicle) by performing routine induction of general anesthesia with propofol 2-3 mg kg-1, fentanyl 1 mcg kg-1. Participants will have mechanical ventilatory support and tidal volume will be set to 8- 10 ml/kg and minute breathing will be set to 16-26. The end tidal carbon dioxide will be kept between 35-40 mmHg. Anesthesia maintenance will be provided with a starting dose of sevoflurane 2% and IV remifentanil 0.05 mcg kg-1 min-1 with a flow of 3 Lt min-1, an Oxygen/air mixture. >20% increase in intraoperative heart rate will be evaluated as pain and remifentanil dose will be increased and the need for remifentanil used intraoperatively will be recorded.

Group ESP (n=30) participants will be given a lateral decubitus position under general anesthesia before the operation and sacral ESP block will be performed accompanied by ultrasound. Group C (n=30) participants who will undergo caudal block will also be given a lateral decubitus position and ultrasound-guided block will be performed.

After 15 minutes of block surgery will be initiated. All operations will be performed by the same experienced team with the same surgical technique.

Near the end of the operation, 15 mg kg-1 IV paracetamol will be given. At the end of the operation, the duration of operation will be recorded.

Pain scoring system Face, Legs, Activity, Cry, Consolability (FLACC) will be recorded in 5th and 30th minutes and 1st, 2nd, 4th, 6th, 12th, 24th hours.

At the end of the operation, the time when there is a need for analgesia will be evaluated as "the first need for analgesia (hour)".

Total amount of additional analgesia (oral paracetamol, mg), amount of rescue analgesia (oral ibuprofen, mg), participants' relative satisfaction (1-Not satisfied, 2-Satisfied, 3-Very satisfied) will be recorded.

Motor weakness, neurological deficit, urinary retention, nausea, vomiting, hypotension, bradycardia, itching, local anesthetic toxicity and bleeding that may occur will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I-II group
* 6 months to 7 years old
* Paediatric age group patients who will undergo hypospadias surgery under general anesthesia

Exclusion Criteria:

* ASA III - IV patient group
* Patients who were operated on urgently
* Patient relatives who did not give consent
* Presence of local anesthetic allergy
* Presence of infection in the area to be blocked
* Presence of coagulation disorder
* Severe organ failure
* Pre-existing neurological deficit
* Mental Retardation
* Anatomical Deformity

Ages: 6 Months to 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 68 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Duration of the analgesia | 1 year
  The duration that elapsed between block application and the patient's first analgesic requirement (if FLACC>3) was evaluated and recorded as ''duration of analgesia (hours)''

SECONDARY OUTCOMES:
Evaluation of the analgesic effects of sacral ESP and caudal block with Face/ Leg/ Activity/ Cry/ Consolability (FLACC) scores in patients undergoing hypospadias surgery. | 1 year
  Evaluation of the analgesic effects of sacral ESP and caudal block with FLACC scores in patients undergoing hypospadias surgery. According to this scoring system, each category is between 0-2, The total score ranges from 0 to 10. 0 points that the game is calm and relaxed, between 1-3 score players are mildly disturbing, scores 4-6 games are moderate He had surgery, scores between 7-10 the player is noticeably disturbing, Pain or harm together reports that
Morphine consumption | 1 year
  Number of patients requiring postoperative morphine, and total postoperative morphine (first 24 hours postoperatively) requirement were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi KESİCİ, Principal Investigator — Sisli Etfal
Locations (1):
- Sisli Hamidiye Etfal Research and Training Hospital, Sarıyer, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mostafa SF, Abdelghany MS, Abdelraheem TM, Abu Elyazed MM. Ultrasound-guided erector spinae plane block for postoperative analgesia in pediatric patients undergoing splenectomy: A prospective randomized controlled trial. Paediatr Anaesth. 2019 Dec;29(12):1201-1207. doi: 10.1111/pan.13758. Epub 2019 Nov 8. PMID 31630465
- [Result] Aksu C, Gurkan Y. Sacral Erector Spinae Plane Block with longitudinal midline approach: Could it be the new era for pediatric postoperative analgesia? J Clin Anesth. 2020 Feb;59:38-39. doi: 10.1016/j.jclinane.2019.06.007. Epub 2019 Jun 13. No abstract available. PMID 31203111
- [Result] Kundra P, Yuvaraj K, Agrawal K, Krishnappa S, Kumar LT. Surgical outcome in children undergoing hypospadias repair under caudal epidural vs penile block. Paediatr Anaesth. 2012 Jul;22(7):707-12. doi: 10.1111/j.1460-9592.2011.03702.x. Epub 2011 Sep 29. PMID 21957982
- [Result] Ozen V, Yigit D. Caudal epidural block versus ultrasound-guided dorsal penile nerve block for pediatric distal hypospadias surgery: A prospective, observational study. J Pediatr Urol. 2020 Aug;16(4):438.e1-438.e8. doi: 10.1016/j.jpurol.2020.05.009. Epub 2020 May 20. PMID 32507565
- [Result] Kaya C, Dost B, Tulgar S. Sacral Erector Spinae Plane Block Provides Surgical Anesthesia in Ambulatory Anorectal Surgery: Two Case Reports. Cureus. 2021 Jan 9;13(1):e12598. doi: 10.7759/cureus.12598. PMID 33585088
- [Result] Topdagi Yilmaz EP, Oral Ahiskalioglu E, Ahiskalioglu A, Tulgar S, Aydin ME, Kumtepe Y. A Novel Multimodal Treatment Method and Pilot Feasibility Study for Vaginismus: Initial Experience With the Combination of Sacral Erector Spinae Plane Block and Progressive Dilatation. Cureus. 2020 Oct 8;12(10):e10846. doi: 10.7759/cureus.10846. PMID 33178502